CLINICAL TRIAL: NCT03620409
Title: Identification of Cardiovascular and Molecular Prognostic Factors for the Mid- and Long-term Outcome of Sepsis
Acronym: ICROS
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: Department of Anesthesiology and Intensive Care Medicine, JUH (Unknown); Department of Cardiothoracic Surgery, JUH (Unknown); Department of Clinical Chemistry and Laboratory Medicine, JUH (Unknown); Department of Biochemistry, Center for Molecular Biomedicine (CMB), FSU Jena (Unknown); Systems Biology and Bioinformatics, Hans-Knöll Institute Jena (Unknown); Institute of Pharmacy, FSU Jena (Unknown)
Responsible Party: Principal Investigator, Sina Coldewey, Principal Investigator, Jena University Hospital
Other Study IDs: ZKSJ106-V1.3; DRKS00013347 (Registry Identifier: DRKS)
Record Dates: First submitted 2018-05-15; First posted 2018-08-08 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Sepsis; Septic Cardiomyopathy; Cardiomyopathies
MeSH Terms: conditions — Sepsis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and stool samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sepsis: Patients with and without diagnosis septic cardiomyopathy Patients with and without suspected or confirmed SARS-CoV-2 infection
- Cardiomyopathy without infection: Patients without operation and patients with scheduled LVAD-Implantation
- Healthy subjects: Healthy controls

SUMMARY:
Sepsis is a life-threatening condition which can affect people of any age. An infection triggers a host response resulting in organ failure. The extent of the organ dysfunction varies between patients and during the course of the condition. Thus far, the only causal treatment option consists in treating the infection early e. g. by an operation or the use of antibiotics. Owing to advances in modern critical care, more patients survive sepsis. Nonetheless, sepsis survivors frequently show impaired organ function, physical disability and considerably decreased health-related quality of life.

It is hypothesized that sepsis-induced cardiac dysfunction - septic cardiomyopathy - may influence mortality. The relationship between occurrence of cardiovascular dysfunction and metabolic changes in the course of sepsis remains unclear. Therefore, the aim of this study is the investigation of cardiovascular function, oxygen consumption and metabolic changes in septic patients. Apart from cardiological routine procedures (echo- and electrocardiography) a newly developed method for measuring the oxygen tension and consumption, bioelectrical impedance analysis for body composition estimation and liver fibrosis assessment via transient elastography will be employed. Through blood, stool and urine analysis, both routine parameters and parameters focusing on patient metabolism will be analysed.

Septic patients will be assessed in the acute phase (3 and 7 days after sepsis diagnosis), the stable phase (at intensive care unit discharge) and after full or incomplete recovery (during two outpatient visits at 6 and 12 months after sepsis diagnosis). The results will be compared with healthy individuals and patients with existing heart disease (cardiomyopathy).

The study aims to identify clinical parameters and signaling pathways involved in the development and course of sepsis. Furthermore, specific parameters associated with the medium- and long-term health status, physical performance and quality of life after sepsis are to be identified. The overall aim of the study is the development of novel diagnostic and therapeutic approaches in sepsis.

DETAILED DESCRIPTION:
The overall aim of the study is the identification of theragnostic targets for the development of novel diagnostic and therapeutic approaches in sepsis. In sepsis, a dysregulated host response to infection leads to organ failure. The extent of organ dysfunction varies between patients and at different stages of the disease. Advances in modern critical care have reduced 28-day mortality over the last years. Nonetheless, a large proportion of sepsis survivors reports long-term physical, mental and cognitive impairments (post intensive care syndrome) including persistent organ dysfunction (persistent critical illness). In addition, mortality rates are considerably increased up to years after sepsis. However, the underlying molecular mechanisms remain unclear.

There is evidence that the development of septic cardiomyopathy may influence mortality. The relationship between the occurrence of cardiovascular dysfunction and metabolic changes in the course of sepsis has not yet been investigated. Therefore, the key aim of this study is the investigation of cardiovascular function, oxygen consumption and metabolic changes in septic patients. Apart from cardiological routine procedures (echo- and electrocardiography) a newly developed method for measuring the mitochondrial oxygen tension and consumption (COMET) will be applied. As oedema is involved in the pathogenesis of altered microcirculation in sepsis, endothelial dysfunction will be analysed via a set of surrogate parameters and body composition (especially extracellular water) measurement via bioelectrical impedance analysis. Liver fibrosis will be assessed via transient elastography. In blood, stool and urine, routine parameters and the metabolome, lipidome and microbiome will be analysed. Septic patients will be assessed in the acute phase (3 and 7 days after sepsis diagnosis), the stable phase (at intensive care unit discharge) and after full or incomplete recovery (during two outpatient visits at 6 and 12 months sepsis diagnosis). Analyses will be complemented by in-depth anamnestic and clinical-epidemiological assessment as well as subsequent information on health related quality of life (EQ-5D-3L) and physical performance (6-minute walk test).

The primary endpoint of the study is the difference in mortality rates between septic patients with and without septic cardiomyopathy six months after sepsis diagnosis. Further research questions include differences in clinical and laboratory parameters between these patient groups during the acute phase, and during the mid-, and long-term course.

The results will be compared with healthy individuals and patients with cardiomyopathy in absence of infection.

ELIGIBILITY:
Inclusion Criteria:

Patients with Sepsis:

* sepsis or septic shock according to Sepsis-3 criteria
* first infection-associated organ dysfunction (= sepsis diagnosis) no older than 72 hours (first blood sample within 96 hours after sepsis diagnosis)
* written informed consent of the patient or his legal representative

Patients with cardiomyopathy without inflammation:

* cardiomyopathy without inflammation
* written informed consent

Healthy subjects:

- written informed consent

Exclusion Criteria:

Patients with sepsis:

* cardiac surgery ≤ 12 months
* sepsis/septic shock ≤ 8 months
* significant pre-existing heart condition

  * endocarditis
  * higher-grade valvular heart disease (grade 3 valve disease, symptomatic aortic stenosis, medium-degree mitral valve insufficiency with reduced ejection fraction or clinical symptoms)
  * complex structural congenital heart disorders (e.g. TGA, Fallot-Tetralogie, endocardial cushion defect)
  * pre-existing significantly reduced cardiac performance (ejection fraction < 45 % or 10 % below norm value)
  * pre-existing pulmonary hypertension
  * myocardial infarction ≤ 1 year in patient history
  * heart transplantation in patient history
  * permanent atrial fibrillation
* pneumectomy in medical history
* contraindication for transesophageal echocardiography (e.g. esophageal resection, higher-grade esophagus varices) and insufficient sonography conditions for transthoracic echocardiography
* liver cirrhosis Child C
* terminal kidney disease with dialysis
* pregnancy/breastfeeding
* previous participation in this study
* participation in another intervention study
* therapy limitation, DNR / DNI order
* life expectancy ≤ 6 months due to comorbidities
* cardiopulmonary resuscitation < 4 weeks before onset of sepsis

Patients with cardiomyopathy without infection:

* sepsis/septic shock ≤ 8 months
* acute organ failure (except cardiac decompensation/cardiogenic shock due to dilated cardiomyopathy) ≤ 6 months due to infection
* complex structural congenital heart disorders (e.g. TGA, Fallot-Tetralogie, endocardial cushion defect)
* infection at point of inclusion
* cardiogenic shock at point of inclusion
* heart transplantation in medical history
* mechanical heart assist device
* pneumonectomy in medical history
* liver cirrhosis Child C
* terminal kidney disease with dialysis
* contraindication for transesophageal echocardiography (e.g. esophageal resection, higher-grade esophagus varices) and insufficient sonographic conditions for transthoracic echocardiography
* pregnancy/breastfeeding
* therapy limitation / DNR / DNI order
* life expectancy ≤ 6 months due to comorbidities
* previous participation in this study
* participation in another interventional study
* cardiopulmonary resuscitation < 4 weeks

Healthy subjects:

* sepsis/septic shock ≤ 8 months
* ICU treatment ≤ 6 months
* infection at point of inclusion
* heart surgery (including heart transplantation) in medical history
* significant pre-existing cardiac condition

  * higher-degree valvular heart disease (grade 3 valve disease, symptomatic aortic stenosis, medium-degree mitral valve insufficiency with reduced ejection fraction or clinical symptoms)
  * complex structural congenital heart disorders (e.g. TGA, Fallot-Tetralogie, endocardial cushion defect)
  * pre-existing significantly reduced cardiac performance (ejection fraction < 45 % or 10 % below norm value)
  * pre-existing pulmonary hypertension
  * myocardial infarction ≤ 1 year in medical history
* pneumonectomy in medical history
* liver cirrhosis Child C
* terminal kidney disease with dialysis
* contraindication for transesophageal echocardiography (e.g. esophageal resection, higher-grade esophagus varices) and insufficient sonography conditions for transthoracic echocardiography
* pregnancy/breastfeeding
* life expectancy ≤ 6 months due to comorbidities
* previous participation in this study
* participation in another intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care and community sample
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Mortality differences between septic patients with vs. without septic cardiomyopathy six months after sepsis diagnosis | Six months after sepsis diagnosis
  Difference in mortality rates between septic patients with vs. without septic cardiomyopathy six months after sepsis diagnosis

SECONDARY OUTCOMES:
Mortality differences between septic patients with vs. without septic cardiomyopathy twelve months after sepsis diagnosis | Twelve months after sepsis diagnosis
  Difference in mortality rates between septic patients with vs. without septic cardiomyopathy twelve months after sepsis diagnosis
Incidence of septic cardiomyopathy | from enrollment until 3 days after ICU discharge
  Estimation of incidence of septic cardiomyopathy in the acute phase of sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Sina M Coldewey, MD, PhD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Jena University Hospital
Locations (1):
- NWG Translational Septomics, Zentrum für Innovationskomepetenz (ZIK) Septomics, Universitätklinikum Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Standke A, Neu C, Baumbach P, Plooij AK, Skitek K, Gotze J, Coldewey SM. Reversible impairment of non-invasively assessed mitochondrial oxygen metabolism in the long-term course of patients with sepsis: a prospective monocentric cohort study. Intensive Care Med Exp. 2025 Nov 14;13(1):114. doi: 10.1186/s40635-025-00808-x. PMID 41233688
- [Derived] Coldewey SM, Neu C, Baumbach P, Scherag A, Goebel B, Ludewig K, Bloos F, Bauer M. Identification of cardiovascular and molecular prognostic factors for the medium-term and long-term outcomes of sepsis (ICROS): protocol for a prospective monocentric cohort study. BMJ Open. 2020 Jun 23;10(6):e036527. doi: 10.1136/bmjopen-2019-036527. PMID 32580988
- See also: Homepage — https://www.septomics.de/en/translational-septomics.html